CLINICAL TRIAL: NCT04778501
Title: Post-market Clinical Follow-Up (PMCF) Study to Investigate Rotational Stability, Visual Outcomes, Contrast Sensitivity, Patient Satisfaction and PCO Rate After Implantation of a Monofocal Toric IOL in an Asian Population
Brief Title: PMCF Study on Monofocal Toric IOL (PODEYE TORIC) in Asia
Acronym: PHY2102
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaver-Visitec International, Inc. (Industry)
Collaborators: targomedGmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHY2102
Record Dates: First submitted 2021-02-24; First posted 2021-03-03 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Cataract; Lens Opacities; Astigmatism
Keywords: Intraocular Lens; Monofocal; Toric Lens
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PODEYE TORIC IOL Implantation experimental (Experimental): Mono- or bilateral implantation of toric intraocular lenses PODEYE TORIC
  Interventions: Device: IOL implantation experimental

INTERVENTIONS:
Device: IOL implantation experimental — Mono- or bilateral implantation of toric intraocular lenses PODEYE TORIC. If only one eye qualifies for toric lens implantation due to small amount of pre-existing corneal astigmatism, one eye will be implanted with PODEYE TORIC and the contralateral eye will be receive an implantation with the monofocal parent lens PODEYE (PhysIOL sa/nv, Liège, Belgium).

SUMMARY:
This is a single-center, prospective, open-label PMCF study whereby patients undergoing routine cataract surgery will have mono- or bilateral implantation of hydrophobic acrylic monofocal toric intraocular lens PODEYE TORIC (study no. PHY2102)

DETAILED DESCRIPTION:
This is a single-center, prospective, open-label PMCF study whereby patients undergoing routine cataract surgery will have mono- or bilateral implantation of hydrophobic acrylic monofocal toric intraocular lens PODEYE TORIC. The device under investigation is a hydrophobic acrylic monofocal toric intraocular lens (IOL) manufactured by the sponsor of this study. The refractive power of the lens has a spherical and a cylindrical component. The IOLs will be implanted in the course of routine cataract surgery and will benefit to patients suffering from cataract development and showing pre-existing corneal astigmatism.

If only one eye qualifies for toric lens implantation due to small amount of pre-existing corneal astigmatism, one eye will be implanted with PODEYE TORIC and the contralateral eye will be received an implantation with the monofocal parent lens PODEYE.

The study purpose is to determine safety, rotational stability, refractive and visual performance, contrast sensitivity, patient satisfaction and PCO rate after mono- or bilateral implantation of PODEYE TORIC intraocular lens.

In total approx. 45 patients will be recruited for this clinical study and undergo mono- or bilateral implantation of PODEYE TORIC intraocular lens. The maximum time between 1st and 2nd eye implantation is 30 days.

Subjects participating in the trial will attend a total of maximum 12 study visits over a period of 330-420 days (preoperative, operative, 1-2 days, 7-14 days, 30-60 days, 120-180 days and 330-420 days postoperative visits). Subjects would have the option for unscheduled visits if required medically.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults ages 50 years or older on the day of screening who have clinically documented cataracts in both eyes;
* Calculated IOL power (sphere and cylinder) is within the range of the investigational IOLs;
* Regular corneal astigmatism (measured by a topographer);
* Corneal astigmatism ≥0.75 D and ≤ 4.25 D (measured by an automatic keratometer) in one or both eyes;
* Capability to understand and sign an IRB approved informed consent form and privacy authorization;
* Clear intraocular media other than cataract;
* Dilated pupil size large enough to visualize IOL axis markings postoperatively;
* Best corrected visual acuity projected to be better than 0.2 logMAR after toric IOL implantation;
* Willing and able to conform to the study requirements.

Exclusion Criteria:

* Age of patient <50 years at the day of screening;
* Regular corneal astigmatism <0.75 D or >4.25 D (measured by an automatic keratometer) in both eyes
* Irregular astigmatism (measured by a topographer);
* Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal or optic disorders);
* Subjects with AMD suspicious eyes as determined by OCT examination;
* Previous intraocular or corneal surgery;
* Traumatic cataract;
* History or presence of macular edema;
* Instability of keratometry or biometry measurements; Acceptable maximum standard deviation: AL: ± 150 µm; ACD: ± 150 µm; K1 / K2: ± 0.15 D;
* Clinically significant, uncontrolled glaucoma with expected negative impact on Contrast Sensitivity and/or visual acuity outcomes;
* Pregnant, lactating or, if able to bear children, unwilling to use medically acceptable birth control over the course of the study;
* Concurrent or previous (within 30 days) participation in another drug or device investigation;
* Clinically significant dry eye as determined by the investigator´s judgement;
* Ocular surface disease (clinical symptoms or keratitis);
* Patients showing contraindications as listed in the current Instructions for use (IFU);
* Unsuitable for study participation for any other reason, as determined by Investigator's clinical judgment (reason to be documented on eCRF).

In addition to above mentioned in- and exclusion criteria, subjects shall be discontinued when certain conditions are present at the time of surgery, including:

* zonular instability;
* need for iris manipulation;
* capsular fibrosis or other opacity; and
* inability to fixate IOL in desired position. In such cases, the subject shall be followed until the condition has stabilized.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Rotational stability - Photograph of IOL with dilated pupil to asses IOL rotation | 6 months postoperative
  The primary performance endpoint is to show statistically non-inferior rotational stability outcomes on PODEYE TORIC lens compared to CER data obtained for a multifocal toric IOL (POD FT) by the same manufacturer sharing the same haptic design but based on a hydrophilic lens material. The null hypothesis is that the absolute mean IOL rotation measured on PODEYE TORIC is not larger than the absolute mean IOL rotation reported in the current CER on POD FT lens.
  The alternative hypothesis is that the absolute mean IOL rotation measured on PODEYE TORIC is larger than the outcomes reported in the current CER on POD FT lens. The measure is taken at 6 months postoperative visit compared to the measurement performed within 10 minutes after surgery.

SECONDARY OUTCOMES:
Best Corrected Distance Visual Acuity compared to historical Data | Pre-Op, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The objective is to compare CDVA above defined thresholds of the investigational product to the results of historical data of EN ISO 11979-7:2018, Annex E (Table E.3 and E.4). The null hypothesis for the CDVA is that / when the true rate of cases with visual acuity 0.3 logMAR or better is less than or equal to the SPE rate. The alternative hypothesis is that the "success" rate is higher than the SPE rate. If the distance corrected visual acuity is 0.3 logMAR or better in 30 eyes or more (with 36 eyes included), the null hypothesis could be rejected, and the alternative hypothesis could be accepted.
Change in cylindrical Power of the Eye | Pre-Op, 1 month postoperative, 6 months postoperative, 12 months postoperative
  Change in cylindrical power, defined as the difference between magnitude of preoperative keratometric cylinder and postoperative manifest cylinder is calculated at every Form. The outcomes of this calculation will be stratified per 0.25D step of preoperative keratometric cylinder and descriptive statistics (mean, standard deviation, median, minimum, maximum) will be provided.

OTHER OUTCOMES:
Intraocular pressure (IOP) measurement | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The IOP will be measured with non-contact tonometer as part of the routine follow up examinations. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Keratometry | Pre-Op, 1 month postoperative, 6 months postoperative
  Keratometric measurements are performed to calculate the required IOL power. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Biometry | Pre-Op
  Biometry measurements are performed to calculate the required IOL power. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
IOL power | during surgery
  The power of the implanted IOL must be recorded.
Target refraction | during surgery
  The target refraction given by the IOL calculator is documented. This parameter is needed to calculate the accuracy of achieving the target refraction. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Fundus OCT | Pre-Op, 6 months postoperative
  An OCT (optical coherence tomography) image will be taken at the preoperative visit to identify AMD suspicious eyes that need to be excluded from this study. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Pupil Size (photopic) | Pre-Op, 6 months postoperative
  Photopic pupil diameters are measured with a precision of at least +/-0.5 mm. For the photopic pupil diameters, eye illumination should be identical to that used for photopic contrast sensitivity testing. It is required that pupil measurements be made with an infrared pupillometer / CCD camera. Pupil measurements should only be made after the eye has had time to fully adapt to the testing conditions (at least 10 minutes).
  The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Pupil Size (mesopic) | Pre-Op, 6 months postoperative
  Mesopic pupil diameters are measured with a precision of at least +/-0.5 mm. For the mesopic pupil diameters, eye illumination should be identical to that used for mesopic contrast sensitivity testing. It is required that pupil measurements be made with an infrared pupillometer / CCD camera. Pupil measurements should only be made after the eye has had time to fully adapt to the testing conditions (at least 10 minutes).
  The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
Manifest refraction | Pre-Op, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The manifested refraction is measured by means of a phoropter. The data contains values for sphere, cylinder and axis of cylinder according to ISO 11979-7:2018.
Uncorrected Distance Visual Acuity (UDVA) - monocular | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions.
Uncorrected Distance Visual Acuity (UDVA) - monocular mesopic | 6 months postoperative, 12 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done monocularly under mesopic conditions.
Uncorrected Distance Visual Acuity (UDVA) - binocular | 6 months postoperative, 12 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions.
Uncorrected Distance Visual Acuity (UDVA) - binocular mesopic | 6 months postoperative, 12 months postoperative
  UDVA is measured with ETDRS charts placed in 4m distance according to ISO 11979-7:2014. This assessment is done binocularly under mesopic conditions.
Corrected Distance Visual Acuity (CDVA) - monocular | Pre-Op, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done monocularly under photopic conditions.
Corrected Distance Visual Acuity (CDVA) - monocular mesopic | 6 months postoperative, 12 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done monocularly under mesopic conditions.
Corrected Distance Visual Acuity (CDVA) - binocular | 6 months postoperative, 12 months postoperative, 24 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done binocularly under photopic conditions.
Corrected Distance Visual Acuity (CDVA) - binocular mesopic | 6 months postoperative, 12 months postoperative
  CDVA is measured with ETDRS charts placed in 4m distance with best aided corrective glasses according to ISO 11979-7:2014. This assessment is done binocularly under mesopic conditions.
Binocular Contrast Sensitivity under photopic light conditions | 6 months postoperative, 12 months postoperative
  Contrast Sensitivity under photopic light conditions using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Binocular Contrast Sensitivity under mesopic light conditions | 6 months postoperative, 12 months postoperative
  Contrast Sensitivity under mesopic light conditions using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Binocular Contrast Sensitivity under photopic light conditions and using a glare source | 6 months postoperative, 12 months postoperative
  Contrast Sensitivity under photopic light conditions with a glare source using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Binocular Contrast Sensitivity under mesopic light conditions and using a glare source | 6 months postoperative, 12 months postoperative
  Contrast Sensitivity under mesopic light conditions with a glare source using the standardized contrast sensitivity device Clinical Trial Suite (M&S Technologies). This examination is performed binocularly.
Patient reported outcomes, Quality of Vision Questionnaire | Pre-Op, 6 months postoperative
  Outcomes measures of a questionnaire to address subjective study outcomes and disturbance by photic phenomena. For this study, the validated and verified questionnaire Quality of Vision (QoV) will be used.
  The QoV Questionnaire consists of a Rasch-tested, linear-scaled, 30-item instrument on three scales providing a QoV score in terms of symptom frequency, severity, and bothersome. It is suitable for measuring QoV in patients with all types of refractive correction, eye surgery, and eye disease that cause QoV problems [McAlinden, 2010]. The score ranges are 0 to 100 with smaller scales indicating better results.
Slitlamp examination - Corneal Status | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Corneal Status
Fundus examination with dilated pupil | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Fundus
Slitlamp examination - Signs of inflammation | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  * Signs of inflammation
  * Anterior chamber cells,
  * Anterior chamber flare,
  * Cystoid macular oedema,
  * Hypopyon, and
  * Endophthalmitis
Slitlamp examination - Pupillary block | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Pupillary block
Slitlamp examination - Retinal detachment | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Retinal detachment
Slitlamp examination - Status of anterior and posterior capsule | Pre-Op, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • Status of anterior and posterior capsule
Slitlamp examination - IOL decentration | 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL decentration
Slitlamp examination - IOL tilt | 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL tilt
Slitlamp examination - IOL discoloration | 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL discoloration
Slitlamp examination - IOL opacity | 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The slitlamp examination is one examination to analyse the integrity of eye structures and the implanted IOL. The examination is performed and documented according to the guidelines in ISO 11979-7:2018.
  With the slitlamp the ophthalmologist can observe the eyes stereoscopically. A focussed slit of light, which can be width-adjusted, is projected on the eye to be examined. The investigator observes this projection on the eye through a reflected light microscope. The slitlamp is used to observe the anterior and posterior part of the eye, including cornea, lens and anterior chamber. By dilating the pupil the fundus can also be examined. Following conditions shall be examined with the slitlamp:
  • IOL opacity
Manual assessment of IOL axis position | within 10 minutes after surgery, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  IOL axis will be subjectively measured by the examiner during the slit lamp examination with dilated eyes. Only for the PODEYE toric implanted eyes.
PCO grading | 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative, 24 months postoperative
  Posterior capsule grading should be performed after pupil dilation at the follow up visits mentioned in the examination matrix. The status of the posterior capsule should be noted to be either "intact" or "not intact". If the capsule is intact, the presence of PCO and/or Elschnig's pearls will be documented as "present" or "absent". If "present", the location and clinical significance of the finding will be documented. Posterior capsular opacification (PCO) will be graded using the following scale:
  0: None
  1. Minimal
  2. Mild
  3. Moderate
  4. Severe
Halo and Glare Scores (binocular) | Pre-Op, 6 months postoperative
  A Halo and Glare simulator software (Eyeland Design Network GmbH, Germany) will be used to assess the subjective perception of photic phenomena. The patients will be asked to adjust the halo and glare level in a simulated image to the amount they perceive of such photic phenomena. This test is performed pre- and postoperatively. The preoperative outcomes serve as a baseline measurement.
  This simulator utilizes a scale for intensity, size of the halo, and glare that ranges from zero (none) to 100 (extremely disturbing). It also allows for classifying the halos into three types, as follows: T1 (diffuse halo ring), T2 (starburst type), and T3 (distinct halo ring) [Kretz, 2015].
Safety outcomes | Pre-Op, during surgery, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  The SPE rates of the investigational product will be compared to the results of historical data of EN ISO 11979-7:2018, Annex E (Table E.2).
  Rates of adverse events as determined by EN ISO 11979-7:2018 will be reported through the complete study follow-up. The proportion of all subjects with these events will be reported over time. Statistical comparisons to EN ISO 11979-7:2018 SPE (Safety and Performance Endpoints) rates (Annex E) will be based on all eyes implanted with the investigational device using a one-sided, exact test based on the binomial distribution.
Medication Revision | Pre-Op, during surgery, 1 day postoperative, 1 week postoperative, 1 month postoperative, 6 months postoperative, 12 months postoperative
  Prior to the study start, a standard medication will be defined that all patients will receive and that is standard for cataract surgery. Only changes to the standard concomitant medication will be documented in the CRFs.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Edward Ang, MD, Principal Investigator — Asian Eye Institute
Locations (1):
- Asian Eye Institute, Makati City, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McAlinden C, Pesudovs K, Moore JE. The development of an instrument to measure quality of vision: the Quality of Vision (QoV) questionnaire. Invest Ophthalmol Vis Sci. 2010 Nov;51(11):5537-45. doi: 10.1167/iovs.10-5341. Epub 2010 May 26. PMID 20505205
- [Background] Kretz FT, Breyer D, Klabe K, Hagen P, Kaymak H, Koss MJ, Gerl M, Mueller M, Gerl RH, Auffarth GU. Clinical Outcomes After Implantation of a Trifocal Toric Intraocular Lens. J Refract Surg. 2015 Aug;31(8):504-10. doi: 10.3928/1081597X-20150622-01. PMID 26274516